CLINICAL TRIAL: NCT01631305
Title: Efficacy and Safety of Levothyroxine in Critical Children With Euthyroid Sick Syndrome in a Pediatric Intensive Care Unit.
Brief Title: Levothyroxine for Children With Euthyroid Sick Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinaloa Pediatric Hospital (Other)
Responsible Party: Principal Investigator, Jesús Javier Martínez-García, Principal investigator, Sinaloa Pediatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HPS-01
Record Dates: First submitted 2012-06-26; First posted 2012-06-29 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Euthyroid Sick Syndrome
Keywords: Euthyroid Sick Syndromes; Thyroxine; Intensive care
MeSH Terms: conditions — Euthyroid Sick Syndromes | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levothyroxine (Experimental): 3 mcg/kg/day
  Interventions: Drug: Levothyroxine
- Control (Placebo Comparator): Calcium magnesia.
  Interventions: Other: Calcium magnesia

INTERVENTIONS:
Drug: Levothyroxine — 3 mcg/kg/day
  Other Names: Brand: Eutirox.
  Arms: Levothyroxine
Other: Calcium magnesia — Placebo.
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether levothyroxine is effective and safe in the treatment of children with euthyroid sick syndrome, hospitalized in a pediatric intensive care unit.

DETAILED DESCRIPTION:
Children with euthyroid sick syndrome, hospitalized in a pediatric intensive care unit, will be randomised to receive either Levothyroxine or placebo, to determine if it diminishes mortality.

ELIGIBILITY:
Inclusion Criteria:

* All children aged 1 month to 17 years.
* Admitted to pediatric intensive care unit.
* TSH and thyroid hormones below age specific levels.

Exclusion Criteria:

* Known thyroid condition.
* Brain death.
* Gut conditions that contraindicate oral route.
* Readmissions to intensive care unit.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
All cause mortality | participants will be followed for the duration of hospital stay, an expected average of 3 weeks

SECONDARY OUTCOMES:
Length of time in intensive care | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Ventilation days | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Use of vasopressors | participants will be followed for the duration of hospital stay, an expected average of 3 weeks
Thyroid hormones levels | participants will be followed for the duration of hospital stay, an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jesus J Martinez, MD, Study Chair — Sinaloa Pediatric Hospital
Locations (1):
- Sinaloa Pediatric Hospital, Culiacán, Sinaloa, Mexico

REFERENCES:
- See also: Sinaloa Pediatric Hospital — http://hospitalpediatrico.org/